CLINICAL TRIAL: NCT00304863
Title: Addition of a Probiotic (Lactobacillus GG) to Metronidazole for the Treatment of Clostridium Difficile Associated Disease
Brief Title: Addition of Lactobacillus to Metronidazole in Treatment of CDAD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The assistant who was going to do this study moved to a different med center
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Daniel M. Musher MD, Principle Investigator, Michael E. DeBakey VA Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-17937
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Enterocolitis; Pseudomembranous Colitis; Antibiotic-associated Colitis
Keywords: CDAD; Clostridium difficile Associated Diarrhea
MeSH Terms: conditions — Enterocolitis; Enterocolitis, Pseudomembranous | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Arm 1 (No Intervention): This are will not receive Lactobacillus
- Arm 2 (Experimental): This arm will receive lactobacillus
  Interventions: Drug: Lactobacillus GG

INTERVENTIONS:
Drug: Lactobacillus GG — This arm will receive the additional probiotic of lactobacillus GG
  Other Names: Lactobacillus
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine whether dietary supplementation with Lactobacillus GG will reduce the rate of failure or relapse following treatment of CDAD with metronidazole.

DETAILED DESCRIPTION:
Clostridium difficile associated disease (CDAD), which nearly always follows antibiotic therapy, has become increasingly common and important in American hospitals, causing substantial morbidity and mortality. Metronidazole is the recommended treatment for this condition. We have recently reported (Clin Infect Dis, June 2005) that treatment with metronidazole is associated with a 22% rate of failure and 28% rate of relapse. No other medication has been shown to be more effective. There is a substantial theory and some limited data to suggest that dietary supplementation with non-pathogenic normal bowel bacteria will benefit these patients. Lactobacillus GG is the best-standardized and the most extensively studied of these agents.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be identified based on the diagnosis of CDAD. This diagnosis is made bases on the presence of diarrhea, fever, abdominal pain and/or leukocytosis together with a positive fecal assay for Clostridium difficile toxin

Exclusion Criteria:

* Patients who are unable to take oral medications and those with underlying gastrointestinal disease or colonostomy will be excluded.
* Patients currently taking penicillins, cephalosporins, quinolones or tetracyclines will be excluded because these drugs are active against Lactobacillus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08-01 (Estimated); Primary Completion 2010-07-31 (Estimated); Study Completion 2010-07-31 (Estimated)

PRIMARY OUTCOMES:
Response to Treatment | less than 10 days
  the time to resolution of diarrhea caused by diarrhea
Stool sample C. diff toxin assay | 30 days after start of medication
  presence of C. diff toxin in stool after 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, M.D., Principal Investigator — Baylor College of Medicine, Houston VA Medical Center
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States